CLINICAL TRIAL: NCT03580486
Title: Investigation of the Psychometric Properties of the Squares Test in Measuring Hand Function in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, research assistant, Gazi University
Other Study IDs: 844
Record Dates: First submitted 2018-06-29; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Hand Function; Squares Test
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's Disease: Parkinson's Disease (Hoehn and Yahr stage 1-4)
  Interventions: Other: The squares test
- Healthy controls: Healthy people
  Interventions: Other: The squares test

INTERVENTIONS:
Other: The squares test — The squares test (ST) originally used in handedness is modified. The ST is a reliable, not time-consuming and easy to administer test for evaluated hand function.

SUMMARY:
The first aim of the present study was to investigate reliability, validity and responsiveness to the minimal clinically important difference, which is defined as the smallest change in score corresponding to clinically meaningful change realized by patient, of the squares test in people with PD.

The second aim of the study is to determine the relationship between hand function and both trunk control and balance in PD population.

DETAILED DESCRIPTION:
At baseline, the ST, Unified Parkinson's Disease Rating Scale (UPDRS), Hoehn and Yahr (H&Y) Scale, Berg Balance Scale (BBS) and Trunk Impairment Scale (TIS) was applied to the PS group when the patients were "on" period. The ST was repeated after seven days from the first application when PD group were "on" period to evaluate its reliability.

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age
* neurologist-diagnosed idiopathic PD (using UK Brain Bank criteria)
* Hoehn & Yahr (H&Y) stages 1 to 4
* Mini-Mental State Examination ≥ 22/30 (literate and with 5 or more years of education) and ≥18/30 (illiterate and with less than 5 years of education)
* living in the community

Exclusion Criteria:

* individuals with other major diseases (e.g., cancer, stroke, epilepsy, dementia, and severe rheumatoid arthritis)
* preexisting disabilities
* visual impairments
* diagnosis of atypical Parkinsonism
* H&Y stage 5
* previous surgical management of PD

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who apply to the Dokuz Eylül University Hospital will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2015-08-17 (Actual); Study Completion 2015-08-17 (Actual)

PRIMARY OUTCOMES:
The Squares Test | 2 minutes
  The Squares Test is used to evaluate hand function.

SECONDARY OUTCOMES:
The Nine-Hole Peg Test | 2 minutes
  The Nine-Hole Peg Test is used to evaluate hand function.
Berg Balance Scale | 15 minutes
  Functional balance performance was assessed with the Berg Balance scale.
Trunk Impairment Scale | 20 minutes
  Trunk control was assessed by the Trunk Impairment Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Söke, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annett M. Five tests of hand skill. Cortex. 1992 Dec;28(4):583-600. doi: 10.1016/s0010-9452(13)80229-8. PMID 1478086
- [Background] Verheyden G, Willems AM, Ooms L, Nieuwboer A. Validity of the trunk impairment scale as a measure of trunk performance in people with Parkinson's disease. Arch Phys Med Rehabil. 2007 Oct;88(10):1304-8. doi: 10.1016/j.apmr.2007.06.772. PMID 17908573
- [Background] Leddy AL, Crowner BE, Earhart GM. Functional gait assessment and balance evaluation system test: reliability, validity, sensitivity, and specificity for identifying individuals with Parkinson disease who fall. Phys Ther. 2011 Jan;91(1):102-13. doi: 10.2522/ptj.20100113. Epub 2010 Nov 11. PMID 21071506
- [Background] Earhart GM, Cavanaugh JT, Ellis T, Ford MP, Foreman KB, Dibble L. The 9-hole PEG test of upper extremity function: average values, test-retest reliability, and factors contributing to performance in people with Parkinson disease. J Neurol Phys Ther. 2011 Dec;35(4):157-63. doi: 10.1097/NPT.0b013e318235da08. PMID 22020457
- [Background] Proud EL, Miller KJ, Bilney B, Balachandran S, McGinley JL, Morris ME. Evaluation of measures of upper limb functioning and disability in people with Parkinson disease: a systematic review. Arch Phys Med Rehabil. 2015 Mar;96(3):540-551.e1. doi: 10.1016/j.apmr.2014.09.016. Epub 2014 Oct 7. PMID 25301441
- [Background] Gebhardt A, Vanbellingen T, Baronti F, Kersten B, Bohlhalter S. Poor dopaminergic response of impaired dexterity in Parkinson's disease: Bradykinesia or limb kinetic apraxia? Mov Disord. 2008 Sep 15;23(12):1701-6. doi: 10.1002/mds.22199. PMID 18649388
- [Background] Foki T, Vanbellingen T, Lungu C, Pirker W, Bohlhalter S, Nyffeler T, Kraemmer J, Haubenberger D, Fischmeister FP, Auff E, Hallett M, Beisteiner R. Limb-kinetic apraxia affects activities of daily living in Parkinson's disease: a multi-center study. Eur J Neurol. 2016 Aug;23(8):1301-7. doi: 10.1111/ene.13021. Epub 2016 May 1. PMID 27132653
- [Background] Gillen G, Boiangiu C, Neuman M, Reinstein R, Schaap Y. Trunk posture affects upper extremity function of adults. Percept Mot Skills. 2007 Apr;104(2):371-80. doi: 10.2466/pms.104.2.371-380. PMID 17566426
- [Background] Schenkman M, Morey M, Kuchibhatla M. Spinal flexibility and balance control among community-dwelling adults with and without Parkinson's disease. J Gerontol A Biol Sci Med Sci. 2000 Aug;55(8):M441-5. doi: 10.1093/gerona/55.8.m441. PMID 10952366